CLINICAL TRIAL: NCT00165854
Title: Study of E7070 Combined With Capecitabine to Determine Efficacy and Recommended Dose of Combination in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-E044-209; 2004-002597-33 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2006-10

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: E7070

SUMMARY:
Part 1: The primary purpose is to determine the recommended dose of E7070 in combination with capecitabine by dose adjustment. Part 2: The primary purpose is to determine the safety and efficacy of the combination in patients with metastatic CRC resistant to 5-fluorouracil and irinotecan.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Histologically or cytologically confirmed solid tumour refractory to standard therapy or for whom no established therapy exists
* Age >= 18 years
* Karnofsky performance status of >= 70%
* Life expectancy of >= 3 months
* Absolute neutrophil count of >= 1.5 × 109/l, platelet count of ³ 100 × 109/l, haemoglobin level of ³ 10 g/dl (>= 6.2 mmol/l) (prior transfusion is permitted)
* Normal hepatic and renal function as defined by serum bilirubin £ 1.5 times the upper limit of normal, ALT and AST £ 2.5 times the upper limit of normal (£ 5 times the upper limit of normal in the presence of hepatic metastases), creatinine clearance ³ 50 ml/min (by Cockroft-Gault formula)
* Male and female patients
* Written informed consent to participate in the study

Part 1 Exclusion Criteria:

* More than two previous courses of documented myelosuppresive chemotherapy (epidermal growth factor targeted therapy does not constitute a course of chemotherapy)
* CNS metastases (a CT or MRI scan should be done if there is a clinical suspicion of CNS metastases)
* Major surgery, chemotherapy or radiation therapy (except palliative) within 4 weeks of treatment start
* Previous investigational cytotoxic treatment for malignant disease within 30 days before the start of the study
* Any treatment with non-oncological investigational drugs within 30 days before the start of the study
* Pregnancy or breast feeding (all women of childbearing potential must have a pregnancy test before inclusion in the study; post-menopausal women must be amenorrhoeic for at least 12 months). Female patients must use adequate contraceptive protection.
* Fertile males not willing to use contraception or whose female partners are not using adequate contraceptive protection
* Uncontrolled infections
* Clinically significant cardiac impairment or unstable ischaemic heart disease including a myocardial infarction within three months of study entry
* History of alcoholism, drug addiction, or any psychiatric or psychological condition which in the opinion of the investigator would impair study compliance
* History of hypersensitivity to sulphonamides
* Prior severe or unexpected reaction to fluoropyrimidine therapy (which may be explained by dihydropyrimidine dehydrogenase deficiency or hypersensitivity to 5-FU)
* Malabsorption syndrome or other condition which may affect absorption of drug
* Concurrent or previous malignancy of a different tumour type within five years of starting the study except for adequately treated non-melanoma skin cancer or cervical intraepithelial neoplasia
* Treatment within two weeks before the start of the study with any of the following: coumarin anti-coagulants, terfenadine, cisapride, cyclosporin, tacrolimus, theophylline, diazepam, sulphonylurea hypoglycaemics, phenytoin, or carbamazepine
* Legal incapacity

Part 2 Inclusion Criteria:

* Ambulant patients with progressive metastatic CRC who have received prior treatment with 5 FU and irinotecan and/or oxaliplatin either as single agents or in combination. Either 5 FU and/or irinotecan and/or oxaliplatin may have been administered in the adjuvant setting or for the treatment of metastatic disease. Patients who have received both 5-FU and irinotecan or oxaliplatin in the adjuvant setting only must have experienced disease recurrence within one year of starting chemotherapy.
* At least one unidimensionally measurable lesion according to the RECIST criteria
* Age ³ 18 years
* Karnofsky performance status of ³ 70%
* Life expectancy of ³ 3 months
* Absolute neutrophil count of ³ 1.5 × 109/l, platelet count of ³ 100 × 109/l, haemoglobin level of ³ 10 g/dl (³ 6.2 mmol/l) (prior transfusion is permitted)
* Normal hepatic and renal function as defined by serum bilirubin £ 1.5 times the upper limit of normal, ALT and AST £ 2.5 times the upper limit of normal (£ 5 times the upper limit of normal in the presence of hepatic metastases), creatinine clearance ³ 50 ml/min (by Cockroft-Gault formula)
* Male and female patients
* Written informed consent to participate in the study

Part 2 Exclusion Criteria:

* Prior chemotherapy other than 5-FU, irinotecan and/or oxaliplatin
* CNS metastases (a CT or MRI scan should be done if there is a clinical suspicion of CNS metastases)
* Major surgery, chemotherapy or radiation therapy (except palliative) within 4 weeks of treatment start
* Previous investigational cytotoxic treatment for malignant disease within 30 days before the start of the study
* Any treatment with non-oncological investigational drugs within 30 days before the start of the study
* Pregnancy or breast feeding (all women of childbearing potential must have a negative pregnancy test before inclusion in the study; post-menopausal women must be amenorrhoeic for at least 12 months). Female patients must use adequate contraceptive protection.
* Fertile males not willing to use contraception or whose female partners are not using adequate contraceptive protection
* Uncontrolled infections
* Clinically significant cardiac impairment or unstable ischaemic heart disease including a myocardial infarction within three months of study start
* History of alcoholism, drug addiction, or any psychiatric or psychological condition which in the opinion of the investigator would impair study compliance
* History of hypersensitivity to sulphonamides
* Prior severe or unexpected reaction to fluoropyrimidine therapy (which may be explained by dihydropyrimidine dehydrogenase deficiency or hypersensitivity to 5-FU)
* Malabsorption syndrome or other condition which may affect absorption of drug
* Concurrent or previous malignancy of a different tumour type within five years of starting the study except for adequately treated non-melanoma skin cancer or cervical intraepithelial neoplasia
* Treatment within two weeks before the start of the study with any of the following: coumarin anti-coagulants, terfenadine, cisapride, cyclosporin, tacrolimus, theophylline, diazepam, sulphonylurea hypoglycaemics, phenytoin, or carbamazepine
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2003-03

PRIMARY OUTCOMES:
To determine the recommended dose of E7070 in combination with capecitabine by dose adjustment;
to determine the safety, tolerability and efficacy (in terms of response rate and progression-free survival) of the combination in patients with metastatic CRC.

SECONDARY OUTCOMES:
Determine the pharmacokinetic profile of capecitabine and E7070 when administered in combination;
measure duration of response and stable disease; to measure median and one year survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, Study Director — Eisai Limited
Locations (4):
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
- Universitätsklinikum der GHS-Essen, Essen, Germany
- Netherlands Cancer Institute, Amsterdam, Netherlands